CLINICAL TRIAL: NCT00949689
Title: Development and Piloting of CBT for Insomnia in Youth With Comorbid Depression
Brief Title: Young Adult and Teen Sleep Study
Acronym: YATSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH082034-01A1 (NIH); NCT00961584 (obsolete NCT alias)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2011-10

CONDITIONS: Depression; Insomnia
Keywords: adolescence; insomnia; depression; sleep problems; cognitive therapy
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy for insomnia and depression (Experimental): cognitive behavioral therapy for insomnia followed by cognitive behavioral therapy for depression
  Interventions: Behavioral: Cognitive Behavioral Therapy for insomnia and depression
- contol (Active Comparator): participants will receive sleep hygiene, time management techniques and cognitive therapy for depression
  Interventions: Behavioral: Cognitive Behavioral Therapy for insomnia and depression

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for insomnia and depression — Experimental arm: Participants will receive sessions of cognitive behavioral treatment for insomnia followed by sessions of cognitive behavior treatment for depression for a total of about 10-12 therapy sessions Control arm: Participants will receive brief sleep hygiene and time management techniques and cognitive behavior treatment for depression for a total of about 10-12 therapy sessions.

SUMMARY:
This study will develop and test a youth cognitive behavioral insomnia intervention to be employed as an adjunct to depression-focused cognitive behavioral treatments. The primary goal of the study is to improve the treatment and prevention of youth depression beyond that achieved with depression-focused pharmacotherapy and psychotherapies. The investigators' ultimate aim in developing this intervention is to enable a series of future outcome trials focused on improving unipolar depression outcomes in youth with comorbid insomnia, by addressing sleep dysfunction. The study will be recruiting from Kaiser Health Plan members in the Portland,Oregon metropolitan area and participants from the Bay Area region of California.

DETAILED DESCRIPTION:
This controlled clinical trial (RCT) will be conducted at the Portland and UC Berkeley sites, directed respectively by Drs. Clarke and Harvey. We are conducting this small RCT at both sites is to establish the feasibility of conducting a fully-powered RCT at multiple sites to be funded by a later, separate R01 application..

Our goal is to enroll 20-30 cases at each of the two sites, for a total of up to 60 youth (30 per study condition). We propose to enroll this modest sample over a 12 month recruitment period. We expect facilitated referrals from several sources, different at each site. In Portland recruitment will be from the 16 HMO pediatric clinics in the Portland metropolitan area. In Berkeley recruitment will come in part from another region of the same HMO, with referrals facilitated by the Kaiser Permanente Department of Research in Oakland, a sister organization to Dr. Clarke's Center for Health Research (CHR) in Kaiser's Northwest region. Referrals will also come from the UBC Psychology Clinic and Dr. Harvey's Sleep and Psychological Disorders Laboratory.

Identified parents and teens will be sent study recruitment letters followed by phone calls to screened for initial eligibility. If the teen appears to be eligible the teen and parent will be scheduled to come to a baseline assessment interview. The baseline assessment is expected to take between 2-3 hours and in appreciation of their time the teen will receive a gift card for $20 and the parent will receive a gift card for $10. If the teen is eligible they will be randomized to either the control arm: sessions in time management and sleep hygiene as well as sessions of cognitive behavioral therapy for depression, or the experimental arm: a combination of CBT therapy sessions for insomnia and depression. Sessions will last from 10-12 weeks. Follow up assessments will be conducted at 12 and 26 weeks for both parent and teen with the same participant incentives as the Baseline. The teen will be asked to wear the ActiGraph watch and keep sleep diary several times throughout their enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 20, living with a parent or guardian.
* English language fluency.
* Meets DSM-IV criteria for either major depression and/or dysthymia Meets Research Diagnostic Criteria (RDC) for insomnia.
* Portland Oregon site participants must be Kaiser Health plan members.

Exclusion Criteria:

* An active, progressive physical illness (e.g., cancer, respiratory disorder) or neurological degenerative disease (e.g., multiple sclerosis) directly related to the onset and course of the sleep disturbance.
* Evidence from clinical diagnosis or report by youth or parent of sleep apnea, restless legs or periodic limb movements during sleep.
* Mental retardation, autism spectrum disorder, or other significantly impairing pervasive developmental disorder.
* Sleep treatment that might confound the interpretation of sleep outcomes.
* Any non-insomnia, non-depressive disorder if the other comorbid condition is clearly the most severe and most impairing of all current diagnoses, and if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed as a function of participating in any stage of this study. Otherwise, we will allow all other comorbid psychiatric conditions (e.g., anxiety, PTSD).

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Depression remission | 2 years

SECONDARY OUTCOMES:
Improved sleep | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gregory N Clarke, PhD, Principal Investigator — Kaiser Permanente; Allison G Harvey, PhD, Study Director — University of California at Berkeley
Locations (2):
- United States (2):
  - University of California at Berkeley, Berkeley, California
  - Kaiser Permanente Center for Health Research, Portland, Oregon

REFERENCES:
- [Derived] Clarke G, McGlinchey EL, Hein K, Gullion CM, Dickerson JF, Leo MC, Harvey AG. Cognitive-behavioral treatment of insomnia and depression in adolescents: A pilot randomized trial. Behav Res Ther. 2015 Jun;69:111-8. doi: 10.1016/j.brat.2015.04.009. Epub 2015 Apr 14. PMID 25917009